CLINICAL TRIAL: NCT07249918
Title: Facilitating the Measurement and Treatment of the Behavioral Symptoms of Dementia (BPSD) and Understanding Caregiver Burden Using Wearable Devices in Rural Taiwan - A Dyadic Feasibility Pilot Study
Brief Title: Feasibility of Wearables in Dementia Care in Rural Taiwan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ta-wei Guu, Consultant Psychiatrist, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH114-REC3-072
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer's Dementia; Neuropsychiatric Symptoms Related to Neurodegenerative Disease; Wearable Devices; Caregiver Burden of People With Dementia; Circadian Rhythm
Keywords: Wearable device; behavioural and psychological symptoms of dementia (BPSD); Sleep; Alzheimer's dementia; Caregiver Burden
MeSH Terms: conditions — Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: single arm dyadic pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Re-Timer (light therapy glasses) (Experimental): an eyewear emitting specific wavelength of green light.
  Interventions: Device: Re-Timer (light therapy glasses)

INTERVENTIONS:
Device: Re-Timer (light therapy glasses) — an eyewear emitting specific wavelength of green light.

SUMMARY:
Taiwan is becoming a super-aged society, and more older adults are living with Alzheimer's disease. Many people with Alzheimer's experience behavioral and psychological symptoms, such as agitation, sleep problems, or mood changes. These symptoms often lower their quality of life and increase stress for their family caregivers.

This study will test two wearable devices in people with Alzheimer's and their caregivers. One device, called Geneactiv, is a wristwatch that tracks daily activity and sleep. The other device, called Re-Timer, is a light therapy eyewear that may help improve sleep and mood. Researchers will look at how easy the devices are to use, whether participants are willing to wear them for several weeks, and whether the light therapy helps reduce sleep problems or caregiver stress.

The study will also compare information from questionnaires with information collected by the devices. The results may help researchers design future studies using wearable tools to better support people living with dementia and their caregivers.

DETAILED DESCRIPTION:
Taiwan is predicted to become a super-aged society, with people older than 65 years accounting for more than 20% of the population. As the prevalence of Alzheimer's dementia (AD) increases with age, the number of people living with AD will continue to rise. Most of these individuals will experience at least one type of behavioral and psychological symptom of dementia (BPSD). These symptoms not only worsen patients' quality of life but also increase caregiver burden, leading to depression, sleep disturbances, and reduced well-being among caregivers themselves.

Currently, questionnaires completed by caregivers are the main tools used to assess and monitor BPSD. Although validated, these questionnaires can only capture cross-sectional information. In a super-aged society where many caregivers are also older adults with cognitive or physical decline, the accuracy of such assessments may be limited. Previous studies, including our research in the United Kingdom, have shown that even patients with late-stage AD can successfully wear a research-grade actigraphy device (Geneactiv) with good compliance. Device-based measurements offer continuous and objective data and can reveal valuable indicators such as the Sleep Regularity Index (SRI), which may predict both cognitive and physical function over time.

Most treatments for BPSD rely on medications, many of which are not specifically approved for this use and may increase the risk of falls or mortality. Non-pharmacological approaches, such as light-based therapy, provide a promising alternative. The Re-Timer device (an eyewear that emits blue-green light) has demonstrated effectiveness in improving sleep and mood in the general population, with a favorable safety profile. If accepted by individuals with dementia and their caregivers, such wearable devices may reduce sleep problems, agitation, and depressive symptoms, thereby improving the overall quality of life for both groups.

To date, very few studies in Taiwan have applied wearable devices to dementia care. This pilot study therefore aims to evaluate the feasibility and acceptability of two wearable technologies, the Geneactiv actigraphy and the Re-Timer light therapy glasses-among people with Alzheimer's dementia and their caregivers. Ten patient and caregiver pairs will be recruited and followed for twelve weeks. Participants will wear the Geneactiv wrist device for eight weeks and the Re-Timer glasses for four weeks. Sleep quality, behavioral symptoms, caregiver burden, and user experience will be assessed through both questionnaires and device data.

The primary goal is to determine whether dementia patients and caregivers can safely and consistently use these devices. Secondary goals include exploring the preliminary effects of Re-Timer on sleep and BPSD, comparing traditional questionnaire results with digital measurements, and establishing a foundation for future large-scale studies to develop digital biomarkers and technology-assisted interventions for dementia care in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* For participants with dementia:

  1. Clinical diagnosis of probable Alzheimer's disease (AD) or mild cognitive impairment (MCI) due to AD, based on established diagnostic criteria.
  2. Presence of at least one prominent behavioral or psychological symptom of dementia (BPSD), including depression, agitation, apathy, or nighttime sleep disturbance.
  3. Prominent is defined as:

     NPI single-item score ≥ 4 (severity × frequency), or NPI-Q severity score ≥ 2, or PSQI total score ≥ 5 (if sleep disturbance is the main symptom).
  4. Stable living arrangement or care environment for at least two weeks before enrollment.
  5. If receiving any pharmacological or non-pharmacological treatments for BPSD, the dosage and frequency must have remained stable for at least two weeks prior to study participation.
  6. Able and willing to provide informed consent; for those lacking decision-making capacity, consent must be obtained from a legally authorized representative.
* For primary caregivers:

  1. Adult primary caregiver of the enrolled participant.
  2. If receiving treatment for caregiver stress, the dosage and frequency must have been stable for at least two weeks before enrollment.
  3. Willing and able to provide informed consent.

Exclusion Criteria:

* Any medical condition that may increase risk during participation, including:

  1. Retinal disease, active use of photosensitizing medications, recent ocular surgery (within 4 weeks), or photosensitivity disorders (e.g., epilepsy).
  2. Unstable physical or mental condition deemed unsuitable by investigators, such as acute delirium or active respiratory infection (including COVID-19)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality (Pittsburgh Sleep Quality Index, PSQI) | baseline to week 12.
  As measured by Pittsburgh Sleep Quality Index (PSQI), a questionnaire providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.
Actigraphy-Derived Sleep and Circadian Rhythm Variables | From enrollment to the end of trial at 8 weeks
  Device-based sleep and circadian rhythm data will be collected via Geneactiv actigraphy and analyzed using the GGIR open-source algorithm. Key variables include:
  * Sleep-related: sleep onset time, wake-up time, total sleep duration (hours), sleep efficiency (%), and wake after sleep onset (WASO, minutes).
  * Circadian-related: light exposure (lux), M5/L5 (activity amplitude), mean sleep midpoint (MSA), intradaily variability (IV), interdaily stability (IS), daytime napping, and Sleep Regularity Index (SRI).
  These will be summarized as descriptive statistics and examined for longitudinal change.
Feasibility and Acceptability of Device-Based Interventions | From enrollment to the end of trial (12 weeks)
  The feasibility, compliance, and satisfaction of using Geneactiv (for measurement) and Re-Timer (for intervention) will be evaluated through qualitative interviews, device adherence data, and the Quebec User Evaluation of Satisfaction with Assistive Technology - Taiwanese version (QUEST-TW).

SECONDARY OUTCOMES:
Caregiver Burden | Baseline to Week 12.
  As measured by Caregiver Burden Inventory (CBI). A 24-item self-report scale assessing five dimensions of caregiver burden (time-dependence, developmental, physical, social, and emotional). The total score ranges from 0 to 96, where higher scores indicate greater burden.
Behavioral and Psychological Symptoms of Dementia (BPSD) | Baseline to Week 12.
  As measured by Neuropsychiatric Inventory Questionnaire (NPI-Q), which evaluates 12 domains of neuropsychiatric symptoms. Each item is rated for severity (0-3) and distress (0-5), producing a total score range of 0-36 for severity and 0-60 for distress, where higher scores indicate greater symptom severity.

OTHER OUTCOMES:
Patient Baseline Characteristics | Baseline (Day 0)
  Includes age (year/month of birth), sex, marital status, education (years), age at AD/MCI diagnosis, time since BPSD onset, smoking and alcohol use, medical/psychiatric comorbidities, and current treatments.
Caregiver Baseline Characteristics | Baseline (Day 0)
  Includes age (year/month of birth), sex, marital status, education (years), smoking and alcohol use, medical/psychiatric comorbidities, and current treatments.
Patient Cognitive Assessment | Baseline (Day 0).
  Cognitive staging assessed using one validated instrument: CDR (0-5), MMSE (0-30), CASI (0-100), or MoCA (0-30). The most recent assessment within 6 months will be used; reassessment performed if decline is suspected.
Caregiver Cognitive Screening (If Applicable) | Baseline (Day 0).
  For older caregivers or those suspected of decline, cognitive screening will be assessed using CDR (0-5), CASI (0-100), MMSE (0-30), or MoCA (0-30). The most recent assessment within 6 months will be used; reassessment performed if decline is suspected.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Beigang Hospital, Beigang, Yunlin, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We will decide if the IPD can be shared before the end of the study.

REFERENCES:
- [Result] Guu TW, Aarsland D, Ffytche D. Light, sleep-wake rhythm, and behavioural and psychological symptoms of dementia in care home patients: Revisiting the sundowning syndrome. Int J Geriatr Psychiatry. 2022 May;37(5):10.1002/gps.5712. doi: 10.1002/gps.5712. PMID 35470491
- [Result] Guu TW, Brem AK, Albertyn CP, Kandangwa P, Aarsland D, Ffytche D. Wrist-worn actigraphy in agitated late-stage dementia patients: A feasibility study on digital inclusion. Alzheimers Dement. 2024 May;20(5):3211-3218. doi: 10.1002/alz.13772. Epub 2024 Mar 18. PMID 38497216